CLINICAL TRIAL: NCT03760848
Title: Study of Potential for Drug Interactions Mediated by CYP3A4 Inhibition With Aramchol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Collaborators: Hammersmith Medicines Research (Other); Analyst Research Laboratories (Other); Alderley Analytical Ltd. (Industry); Diamond Pharma Services Regulatory Affairs Consultancy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Aramchol 016
Record Dates: First submitted 2018-11-22; First posted 2018-11-30 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-02

CONDITIONS: Healthy
MeSH Terms: interventions — aramchol; Midazolam; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Midazolam, Atorvastatin / Aramchol, Midazolam, Atorvastatin (Other): Midazolam 2 mg -atorvastatin 40 mg /Aramchol 600mg -midazolam 2 mg-atorvastatin 40 mg (MA/MAA)
  Interventions: Drug: Aramchol; Drug: Midazolam; Drug: Atorvastatin

INTERVENTIONS:
Drug: Aramchol — Aramchol 600 mg
Drug: Midazolam — Midazolam 2 mg
Drug: Atorvastatin — atorvastatin 40 mg

SUMMARY:
The trial is an open-label, 2-period, single-sequence assessment of CYP3A4 inhibition by aramchol using the probe substrates midazolam and atorvastatin to assess CYP3A4 activity.

DETAILED DESCRIPTION:
Enrolment of 16 subjects is planned. Each subject will take part in 2 study periods.

In Period 1, subjects will receive a single oral dose of 2 mg midazolam on Day 1 and a single oral dose of 40 mg atorvastatin on Day 3.

In Period 2, subjects will receive twice-daily oral doses of 300 mg aramchol (the IMP) for 18 days. During aramchol dosing, subjects will take a single dose of 2 mg midazolam in the morning on Day 10 and 40 mg atorvastatin in the morning on Day 12.

Subjects will be screened within 21 days before their first dose of study medicine. In Period 1, they will remain resident on the ward from Day -1 to Day 10. In Period 2, subjects will be admitted on Day -1 and discharged on Day 19. Subjects will attend a follow-up visit approximately 2 weeks later, on Day 33 (±2 days). There will be an interval of at least 1 day between Periods 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male healthy volunteers.
2. Aged 18-45 years at time of consent.
3. A body mass index (BMI; Quetelet index) in the range 18.0-30.9.
4. Ability to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of the entire trial.
5. Willingness to give written consent to participate after reading and understanding the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.
6. Agree to use effective contraception as described in section 9.
7. Agree not to donate blood or blood products during the study and for up to 3 months after the administration of the trial medication.
8. Willingness to give written consent to have data entered into The Overvolunteering Prevention System (TOPS).

Exclusion Criteria:

1. Volunteers of East Asian descent including, but not limited to, Chinese, Japanese, Korean, Mongolian, and/or Vietnamese
2. Be a smoker, or have smoked cigarettes or other tobacco or nicotine products in the last 12 months.
3. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or alkaline phosphatase (AP) > Upper Limit of Normal (ULN) at the screening visit. A repeat is allowed on one occasion for determination of eligibility.
5. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous,
6. Presence or history of obstructive sleep apnoea.
7. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs including gastrointestinal disorder or of oesophageal, gastric, biliary or intestinal surgery (excluding herniotomy and appendectomy).
8. Use of anticholinergic or other drugs known to affect gastrointestinal motility during the 7 days before the first dose of trial medication.
9. Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
10. Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines.
11. Presence or history of severe adverse reaction to any drug or a history of sensitivity to aramchol, midazolam or atorvastatin, or any excipients in the tablets.
12. Use of a prescription medicine or any other medicine or herbal remedy (such as St John's wort) during the 28 days before the first dose of trial medication or use of any other over-the-counter medicine, with the exception of acetaminophen (paracetamol), during the 7 days before the first dose of trial medication.
13. Receipt of an investigational product (including prescription medicines) as part of another clinical trial within the 3 months before first admission to this study; in the follow-up period of another clinical trial at the time of screening for this study.
14. Presence or history of drug or alcohol abuse, or intake of more than 14 units of alcohol weekly.
15. Blood pressure and heart rate in supine position at the screening examination outside the ranges: blood pressure 100-140 mm Hg systolic, 50-90 mm Hg diastolic; heart rate 45_90 beats/min, unless judged not clinically significant.
16. Possibility that the volunteer will not cooperate with the requirements of the protocol.
17. Evidence of drug abuse on urine testing.
18. Positive test for hepatitis B, hepatitis C or HIV.
19. Loss of more than 400 mL blood during the 3 months before the trial, eg as a blood donor.
20. Objection by General Practitioner (GP) to volunteer entering trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Midazolam - cmax | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
  Maximum plasma concentration
Atorvastatin - cmax | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
  Maximum plasma concentration
Midazolam - tmax | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
  Time of maximum plasma concentration
Atorvastatin - tmax | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
  Time of maximum plasma concentration
Midazolam - Area under the concentration-time curve to last measurable concentration (AUClast) | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
Atorvastatin - Area under the concentration-time curve to last measurable concentration (AUClast) | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
Midazolam - Area under the concentration-time curve extrapolated to infinite time (AUCinf) | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
Atorvastatin - Area under the concentration-time curve extrapolated to infinite time (AUCinf) | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
Midazolam - %AUCextrapinf | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
  Percentage of AUC that was extrapolated
Atorvastatin - %AUCextrapinf | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
  Percentage of AUC that was extrapolated
Midazolam - t½ | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
  Terminal elimination half-life
Atorvastatin - t½ | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
  Terminal elimination half-life
Midazolam - CL/F | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
  Clearance/fraction of dose absorbed
Atorvastatin - CL/F | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
  Clearance/fraction of dose absorbed
Midazolam - VZ/F | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
  Volume of distribution/fraction of dose absorbed
Atorvastatin - VZ/F | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
  Volume of distribution/fraction of dose absorbed
Midazolam - MRT | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
  Mean residence time
Atorvastatin - MRT | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
  Mean residence time
Midazolam - λz | Blood samples for assay of midazolam will be taken before, and frequently up to 48 hours after each dose.
  Terminal rate constant
Atorvastatin - λz | Blood samples for assay of atorvastatin will be taken before, and frequently up to 168 hours after each dose.
  Terminal rate constant

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, M.D., Principal Investigator — HMR
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No